CLINICAL TRIAL: NCT03098459
Title: Illuminating Neuropsychological Dysfunction and Systemic Inflammatory Mechanisms Gleaned After Hospitalization in Trauma-ICU Study
Acronym: INSIGHT-ICU
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Mayur Patel, Professor, Vanderbilt University Medical Center
Other Study IDs: 171335; R01GM120484 (NIH)
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Delirium; Cognitive Impairment; Alzheimer; Early Onset; Trauma; Polytrauma; Traumatic Brain Injury; ICU; Critical Illness
Keywords: Delirium; Cognitive Impairment; Alzheimer's Disease; Encephalopathy; Trauma; Polytrauma; ICU; Critical Illness; Traumatic Brain Injury; INSIGHT-ICU; INSIGHT; Intracerebral hemorrhage; Subarachnoid hemorrhage; Neurotrauma; Neuropsychology; Dementia; Critical Care; Subdural hemorrhage; Cognition; Neuropsychological Outcomes; Neuropsychology Dysfunction; Inflammation; Neuroinflammation; Inflammatory Mechanisms; Burn; Critically Injured; Injury; Head Injury; Long-term Cognitive Impairment; ICU-related Dementia; Employment; Return to Work
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Alzheimer Disease; Wounds and Injuries; Multiple Trauma; Brain Injuries, Traumatic; Critical Illness; Brain Diseases; Cerebral Hemorrhage; Subarachnoid Hemorrhage; Dementia; Hematoma, Subdural; Inflammation; Neuroinflammatory Diseases; Burns; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically Ill Trauma Patients: Non-intervention observational prospective cohort study
  Interventions: Other: Non-interventional observational prospective cohort study

INTERVENTIONS:
Other: Non-interventional observational prospective cohort study — Non-interventional observational prospective cohort study

SUMMARY:
Cognitive skills are essential to live independently, manage finances, maintain employment, and function in society. Loss of these cognitive skills puts a tremendous burden on society as seen with dementias, Alzheimer's disease, and traumatic brain injury. The INSIGHT-ICU Study (Illuminating Neuropsychological dysfunction and Systemic Inflammatory mechanisms Gleaned after Hospitalization in Trauma-ICU Study) is the first comprehensive and longitudinal long-term cognitive impairment study after traumatic injury. The societal impact of long-term cognitive impairment after trauma is immense given that these patients are young and constitute a large proportion of employable adults.

DETAILED DESCRIPTION:
Cognitive skills are the crucial abilities required to manage money, maintain employment, and live independently. Long-term cognitive impairment (LTCI) is a disabling loss of these skills that can persist for months to years. LTCI frequently occurs after primary brain injury (e.g., traumatic brain injury, hypoxia), but older LTCI research has not characterized primary brain injury using NIH Common Data Elements in Imaging, the contributions of polytrauma, and the time-course of the critical illness, including secondary brain injury (i.e., delirium). In our recent large study of ICU patients without primary brain injury, over 50% of patients had LTCI and nearly 50% were newly unemployed at one-year post-discharge. In-hospital delirium was the major independent risk factor for LTCI. Surprisingly, this delirium-related LTCI was similar to the LTCI seen in past studies after moderate traumatic brain injury. Thus, both primary and secondary brain injury are associated with LTCI, yet they have not been studied together. There is an unmet need to define the independent risks of primary brain injury and delirium in LTCI. The trauma ICU patient is at combined risk for primary brain and/or multisystem injuries, secondary brain injury, and critical illness; these critically injured patients are the unique population to address this knowledge gap.

Therefore, our FIRST HYPOTHESIS is that delirium duration is an independent risk for the severity of LTCI, controlling for confounders of co-morbidities, socioeconomic status, pre-injury employment, primary brain injury, polytrauma, and critical illness. AIM 1 will address this hypothesis by defining the independent risks of primary and secondary brain injury on the severity of LTCI among trauma ICU subjects.

But, LTCI's real-world impact on employment has not been explained or adjusted for the above confounders and social factors. Accordingly, our SECOND HYPOTHESIS is that LTCI severity is an independent risk for lower level of employment, adjusting for similar confounders. AIM 2 will delineate the independent risk of LTCI severity on employment among trauma ICU survivors. Lastly, LTCI pathogenesis may be related to persistent inflammation.

So, our THIRD HYPOTHESIS is that hospital discharge biomarkers of persistent inflammation will be independent risks for LTCI severity, adjusting for similar confounders. AIM 3 will explore the mechanistic role of plasma inflammatory biomarkers on LTCI severity among trauma ICU survivors.

ELIGIBILITY:
Inclusion Criteria:

• Adult trauma and/or burn patients, injury from any mechanism, requiring admission to an Adult ICU for the treatment of shock (any type), respiratory failure, and/or neurologic failure, including monitoring for deteriorating brain function.

Exclusion Criteria:

* Inability to obtain informed consent within the 72 hours following injury

  * Attending physician refusal
  * Patient and/or surrogate refusal
  * 72-hour period of eligibility was exceeded before the patient was screened
  * Patient unable to consent and no surrogate available within the 72-hour period
* Residence > 200 miles from study site and do not regularly visit the Nashville area.
* Patients who are homeless and have no secondary contact person available.
* Severe prior cognitive or neurodegenerative disorder that prevents a patient from living independently at baseline
* Inability to understand English or Spanish or bilateral deafness or bilateral vision loss
* Inability to co-enroll with other studies
* Prisoners
* Substance abuse requiring treatment, known psychotic disorder (e.g., schizophrenia or schizoaffective disorder), or recent (within the past 6 months) serious suicidal gesture necessitating hospitalization
* Expected death within 24 hours of enrollment or lack of commitment to aggressive treatment by family or the medical team (e.g., likely to withdraw life support measures within 24 hours of screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be broadly eligible for inclusion if they are Adult trauma and/or burn patients, injury from any mechanism, requiring admission to an Adult ICU for the treatment of shock (any type), respiratory failure, and/or neurologic failure, including monitoring for deteriorating brain function.
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
LTCI (Long-term Cognitive Impairment) as measured by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 12 months
  LTCI (Long-term Cognitive Impairment) as measured by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)

CONTACTS AND LOCATIONS:
Overall Officials: Mayur B Patel, MD,MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH RePORTER — https://reporter.nih.gov/project-details/9260624